CLINICAL TRIAL: NCT05473130
Title: Breethe Abiomed Recovery RegisTry (BART)
Acronym: BART
Status: Completed | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11202020
Record Dates: First submitted 2022-02-15; First posted 2022-07-25 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-07

CONDITIONS: Cardiopulmonary Bypass; ARDS; Heart Failure
Keywords: Breethe Oxy-1 System; Extracorporeal Membrane Oxygenation; Cardiopulmonary bypass; ARDS; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Breethe Oxy-1 System — To pump, oxygenate, and remove carbon dioxide from blood during cardiopulmonary bypass with Breethe Oxy-1 System

SUMMARY:
The BART Registry intended to utilize observational data of the Abiomed Breethe OXY-1 System™ in real-world settings to drive best practice usage patterns, serve as a tool to measure and improve the quality of patient care and as a resource to inform us on the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* all adult subjects supported with Breethe Oxy-1 System

Exclusion Criteria:

* subjects under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects supported with Breethe Oxy-1 System
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Survival up to the hospital discharge | Up to the hospital discharge, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - AdventHealth Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Maryland, College Park, Maryland
  - NYU School of Medicine, New York, New York
  - UPenn Health System, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No